CLINICAL TRIAL: NCT01743014
Title: A Prospective, Randomized, Two Period, With an Intermediate Wash Out Period, Cross-over Study to Compare the Effects of Either Combined Therapy With Ramipril and Clopidogrel or Ramipril Monotherapy on Oxidative Stress, Vascular Inflammation and Endothelial Dysfunction in Patients With Type 2 Diabetes and Diabetic Nephropathy
Brief Title: Ramipril and Clopidogrel in Oxidative Stress, Vascular Inflammation and Endothelial Dysfunction in Type 2 Diabetes and Diabetic Nephropathy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: AHEPA University Hospital (Other)
Collaborators: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Vaia Bougatsa, Medical Doctor-Resident of Internal Medicine, AHEPA University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 15/10-7-2012
Record Dates: First submitted 2012-11-21; First posted 2012-12-06 (Estimated); Last update posted 2012-12-06 (Estimated); Status verified 2012-11

CONDITIONS: Diabetes Type 2; Diabetic Nephropathy; Vascular Disease
Keywords: diabetes; diabetic nephropathy; vascular inflammation; oxidative stress; endothelial dysfunction; Asymmetric dimethylarginine; High sensitivity CRP; albumine to creatinine ratio; isoprostane; clopidogrel; ramipril; carotid intima media thickness
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetic Nephropathies; Vascular Diseases; Diabetes Mellitus | interventions — Ramipril; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ramipril (Active Comparator): Ramipril 10 mg tablets. Each dose will be taken orally with water once daily.
  Interventions: Drug: Ramipril
- clopidogrel and ramipril (Active Comparator): clopidogrel 75mg tablet and ramipril 10mg. Each drug will be taken orally with water once daily
  Interventions: Drug: Ramipril; Drug: Clopidogrel

INTERVENTIONS:
Drug: Ramipril — Patients will receive 10 mg ramipril throughout the study. Each dose will be taken orally once daily. The duration of treatment with ramipril is 26 weeks
  Other Names: Triatec
Drug: Clopidogrel — 12 weeks treatment with ramipril 10 mg and clopidogrel 75 mg once daily followed by a 2 week wash out period for clopidogrel and subsequently additional 12 weeks treatment wit both drugs after cross over.
  Other Names: Plavix; Iscover
  Arms: clopidogrel and ramipril

SUMMARY:
The purpose of this study is to determine whether the combination with ramipril and clopidogrel leads to further improvement of endothelial function, reduction of oxidative stress and reduction of vascular inflammation, compared with ramipril monotherapy, in patients with Diabetes Mellitus type 2 and diabetic nephropathy.

DETAILED DESCRIPTION:
* Cardiovascular disease is the leading cause of deaths in diabetic population with diabetic nephropathy.
* Pharmacologic therapy for patients with diabetes and hypertension should be with a regimen that includes either an angiotensin-converting-enzyme inhibitor (ACEi) or an angiotensin receptor blocker (ARB)
* Diabetic patients at increased cardiovascular risk should receive an antiplatelet agent for primary prevention.

Methods:

An open label,randomized, two period cross-over design study, involving patients with type 2 diabetes and diabetic nephropathy. After a 4 weeks wash out period for ACE inhibitors or Angiotensin receptor blockers (week 0, baseline) 60 patients will be randomized to receive ramipril(10 mg) only or ramipril (10 mg) and clopidogrel (75mg) for 12 weeks exchanging their treatment for a further 12 weeks, after a 2 week wash out period for clopidogrel. Patients will be examined and measurements will be taken at baseline (week 0), and at the end of 12, 14, and 26 weeks.

ELIGIBILITY:
Inclusion Criteria: type 2 diabetes patients with diabetic nephropathy in the range of micro- or macroalbuminuria and

* HbA1c(glycosylated haemoglobin A1c <7%
* Blood pressure ≤130/80 mmHg
* LDL (Low Density Lipoproteins) <100 mg/dl
* Informed consent

Exclusion Criteria:

* patients with diabetic nephropathy and estimated GFR <30ml/min with Modification of Diet in Renal Disease equation (MDRD equation)
* baseline potassium > 5.2 meq/L
* patients with nephrotic proteinuria defined as albumine to creatinine ratio (ACR)> 3.5 g/g or as proteinuria >3.5 g per 1.73 m2 per 24 hours
* history or evidence of non-diabetic kidney disease
* history of stroke, peripheral artery disease, coronary artery disease
* history or evidence of a secondary form of hypertension
* history of severe hepatic failure, malignancy, severe endocrinopathy,autoimmune disease or chronic inflammatory disease
* any known bleeding or platelet disorder or platelets <100.000/μL
* heart failure in New York Heart Association(NYHA) functional class II-IV
* inability or unwillingness on the part of the patient to sign the Patient Consent Form
* known hypersensitivity to ramipril or to clopidogrel
* Women of child-bearing potential
* use of oral anticoagulants or other antithrombotic treatment
* use of glitazones
* patients receiving statins should be on a stable dose of at least 3 months prior to study initiation and dose should be constant during the study
* any surgical or medical condition which in the opinion of the investigator may expose the patient to a higher risk in participation in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-07; Primary Completion 2014-07 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Changes in Asymmetric dimethylarginine (ADMA) blood levels after the combined treatment with ramipril and clopidogrel compared with ramipril monotherapy | Baseline to week 12 and week 14 to week 26
  The primary aim is to investigate the effect of the combined treatment with ramipril and clopidogrel versus ramipril monotherapy in ADMA as biomarker of endothelial dysfunction.
Changes in High-sensitivity C-reactive protein (HsCRP) blood levels after the combined treatment with ramipril and clopidogrel compared with ramipril monotherapy | Baseline to week 12 and week 14 to week 26
  The primary aim is to investigate the effect of the combined treatment with ramipril and clopidogrel versus ramipril monotherapy in hsCRP as biomarker of vascular inflammation
Changes in soluble CD40 Ligand (sCD40L)blood levels after the combined treatment with ramipril and clopidogrel compared with ramipril monotherapy | Baseline to week 12 and week 14 to week 26
  The primary aim is to investigate the effect of the combined treatment with ramipril and clopidogrel versus ramipril monotherapy in soluble CD40 Ligand as biomarker of vascular inflammation.
Changes in urine 8-isoprostane-F2 levels after the combined treatment with ramipril and clopidogrel compared with ramipril monotherapy | Baseline to week 12 and week 14 to week 26
  The primary aim is to investigate the effect of the combined treatment with ramipril and clopidogrel versus ramipril monotherapy in urine 8-isoprostane-F2 as biomarker of oxidative stress.
Reduction in albumine to creatine ratio after the combined treatment with ramipril and clopidogrel compared with ramipril monotherapy | Baseline to week 12 and week 14 to week 26
  The primary aim is to investigate the effect of the combined treatment with ramipril and clopidogrel versus ramipril monotherapy in albumine to creatine ratio as an index of cardiovascular disease

SECONDARY OUTCOMES:
Changes in ADMA blood levels after treatment with ramipril | baseline to week 26
  Evaluation of the effect of ramipril, as antihypertensive therapy, in endothelial dysfunction in patients with diabetes mellitus type 2 and diabetic nephropathy
Increase of Glomerular Filtration Rate (GFR) after combined treatment with ramipril and clopidogrel and after ramipril monotherapy | baseline to week 12 and week 14 to week 26
Change from baseline in carotid intima-media thickness after combined therapy with ramipril and clopidogrel and after ramipril monotherapy | baselibe to week 12 and week 14 to week 26

CONTACTS AND LOCATIONS:
Overall Officials: Fotios S Iliadis, Lecturer of Internal Medicine, Study Director — AHEPA University Hospital/ Aristotle University of Thessaloniki; Vaia F Bougatsa, Resident of Internal Medicine, Principal Investigator — AHEPA University Hospital/ Aristotle University of Thessaloniki
Locations (2):
- Greece (2):
  - AHEPA University Hospital, Thessaloniki, Thessaloniki
  - Aristotle University of Thessaloniki/ AHEPA University Hospital, Thessaloniki, Thessaloniki

REFERENCES:
- [Derived] Natale P, Palmer SC, Saglimbene VM, Ruospo M, Razavian M, Craig JC, Jardine MJ, Webster AC, Strippoli GF. Antiplatelet agents for chronic kidney disease. Cochrane Database Syst Rev. 2022 Feb 28;2(2):CD008834. doi: 10.1002/14651858.CD008834.pub4. PMID 35224730